CLINICAL TRIAL: NCT06848140
Title: Using High Definition Transcranial Direct Current Stimulation to Treat Verbal Retrieval Deficits Secondary to Chronic Traumatic Brain Injury (STIM-CTBI)
Brief Title: Using Non-invasive Brain Stimulation to Treat Word Finding Difficulty in Chronic Traumatic Brain Injury
Acronym: STIM-CTBI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Hsueh-Sheng Chiang, Assistant Professor, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2025P000171; 4R00DC020185-03 (NIH)
Record Dates: First submitted 2025-02-21; First posted 2025-02-26 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Traumatic Brain Injury; Word Finding Difficulty; Cognitive Symptom; Cognitive Change; Acquired Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic; Anomia; Neurobehavioral Manifestations; Brain Injuries | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: The participants will be randomly assigned to 1 of 2 treatment arms: (1) 1 milliamp transcranial direct current stimulation (tDCS) active treatment applied to pre-supplementary motor area for 20 minutes over 10 sessions to (2) sham tDCS following the same schedule.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants, assessors, and technicians interacting with participants will be blind to assigned conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Active to Sham Transcranial direct current stimulation (Experimental): Subjects in this arm will first be randomly assigned to receive active stimulation. After completion of active stimulation, subjects will be assigned to sham stimulation.
  Interventions: Device: Active Transcranial direct current stimulation; Device: Sham Transcranial direct current stimulation
- Sham to Active transcranial direct current stimulation (Experimental): Subjects in this arm will first be randomly assigned to receive sham stimulation. After completion of sham stimulation, subjects will be assigned to active stimulation.
  Interventions: Device: Active Transcranial direct current stimulation; Device: Sham Transcranial direct current stimulation

INTERVENTIONS:
Device: Active Transcranial direct current stimulation — Transcranial direct current stimulation will be delivered via a Neuroelectrics Starstim 20 or 32. Stimulation will consist of 1 milliamp stimulation, with anodal stimulation delivered at electrode Fz (International 10/10 System for electroencephalography electrode placement) and electrodes F7, FP1, FP2, and F8 as returns. All electrodes are 1 cm diameter Ag/AgCl electrodes and make contact with the scalp via connective gel. Stimulation will linearly ramp up from 0 milliamps to 1 milliamp over 60 seconds, then remain at 1 milliamp of stimulation over 20 minutes, and finally ramping down at to 0 milliamps over 60 seconds.
  Other Names: tDCS; 1 milliamp tDCS; High definition tDCS; High definition transcranial direct current stimulator, Neuroelectrics Starstim 20 or 32
Device: Sham Transcranial direct current stimulation — Sham transcranial direct current stimulation will be delivered via a Neuroelectrics Starstim 20 or 32. The sham setup will consist of anodal electrode Fz (International 10/10 System for electroencephalography electrode placement) and electrodes F7, FP1, FP2, and F8 as returns. All electrodes are 1 cm diameter Ag/AgCl electrodes and make contact with the scalp via connective gel. Stimulation will linearly ramp up from 0 milliamps to 1 milliamp over 60 seconds, ramp down to 0 milliamps over 60 seconds and then be left off for 20 minutes.

SUMMARY:
The purpose of this study is to learn more about how brain stimulation affects word finding problems in people who have a traumatic brain injury (TBI). The type of brain stimulation used is called transcranial direct current stimulation (tDCS). tDCS delivers low levels of electric current to the brain and high definition tDCS (HD-tDCS) delivers the current with multiple electrodes on the scalp. This current is delivered with HD-tDCS to parts of the brain that may help with remembering things. The investigators hope that this can help to improve word finding and memory problems in people with TBI.

DETAILED DESCRIPTION:
The investigators plan to recruit English-speaking participants aged 18-85 years with a history of chronic TBI (> 1 year since injury prior to enrollment), all of whom have problems with cognition. The participants will be randomized to receive (1) active first followed by sham HD-tDCS condition, or (2) sham first followed by active condition in order to assess the efficacy of HD-tDCS on improving verbal retrieval function. The randomization will be double-blinded to the participants and the research personnel who administer the procedures. The study therefore adopts a double-blind randomized cross-over design. The proposed study will measure response to HD-tDCS treatment over the pre-supplementary motor area (preSMA) region when compared to sham with verbal retrieval function (verbal fluency, naming, verbal learning) as the primary outcome. Secondary outcome measures include cognitive performance other than verbal retrieval function and electroencephalography (EEG) measures. The participants will receive two phases of 10 sessions of active stimulation (1 mA anodal HD-tDCS targeting preSMA for 20 min) or sham across 2 weeks. All participants will be blinded to their condition. EEG and neuropsychological tasks will be completed at baseline, immediate follow-up after session 10, and a 2-month follow-up. The participants will also undergo an MRI session at baseline. Those participants randomized into the active or sham group will have the opportunity to return after 2 months and receive sham (if active first) or active (if sham first) treatment and will undergo the EEG and neuropsychological tests again immediately following the last HD-tDCS session and at a 2-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 85
* Fluent in speaking and reading English
* Able to provide informed consent
* Has a TBI at least one year prior to enrollment and not related to military experience
* Has a confirmation of verbal retrieval difficulties as measured by the Verbal Retrieval Difficulty Interview questions

Exclusion Criteria:

* Lifetime major or active neurologic conditions (e.g., stroke, epilepsy, brain tumor, dementia, seizure occurrence less than one year ago)
* Lifetime major or active cardiovascular conditions (e.g., cardiac arrythmia, heart failure, heart attack)
* Current substance use disorder
* Lifetime major psychiatric disorders (e.g., schizophrenia, bipolar disorder)
* Severe depression at the time of enrollment (BDI-II >= 29) or psychiatric ER visits or hospitalization less than 6 months ago prior to enrollment
* Current sensory (e.g., blind, deaf) or physical (e.g., severe motor weakness) impairment that interferes with testing
* Contraindications for tDCS or MRI
* The person cannot be left alone for 8+ hours.
* Not verbally communicative.
* Currently undergoing and not wishing to discontinue speech and cognitive therapy during study participation.
* Incapable of understanding the consent or unable to consent for oneself.
* Unable to travel to BIDMC's Berenson-Allen Center
* Pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
The Controlled Oral Word Association Test - letter fluency | Treatment differences (active versus sham) in change from Baseline to immediately and 2-months Post-Treatment.
  Evaluation of treatment differences (active versus sham) in change on the Control Word Association Test. Metric: Number of Correct Items Generated
The Controlled Oral Word Association Test - category fluency | Treatment differences (active versus sham) in change from Baseline to immediately and 2-months Post-Treatment.
  Evaluation of treatment differences (active versus sham) in change on Category Fluency. Metric: Number of Correct Items Generated
The Boston Naming Test | Treatment differences (active versus sham) in change from Baseline to immediately and 2-months Post-Treatment.
  Evaluation of treatment differences (active versus sham) in change on The Boston Naming Test. Metric: Number of Correct Items Generated.
The Delis Kaplan Color Word Interference Test | Treatment differences (active versus sham) in change from Baseline to immediately and 2-months Post-Treatment.
  Evaluation of treatment differences (active versus sham) in change on the Delis Kaplan Color Word Interference Test. Metric: Time to Name Items
Rey Auditory Verbal Learning Test and alternative lists | Treatment differences (active versus sham) in change from Baseline to immediately and 2-months Post-Treatment.
  Evaluation of treatment differences (active versus sham) in change in Rey Auditory Verbal Learning Test. Metric: Number of Total learning items and Correct Recalls.

SECONDARY OUTCOMES:
The Trail Making Test (Parts A & B) | Treatment differences (active versus sham) in change from Baseline to immediately and 2-months Post-Treatment.
  Evaluation of treatment differences (active versus sham) in change on the Trail Making Test (Parts A&B). Metric: Time to Solution
Digit Span Forward & Backward | Treatment differences (active versus sham) in change from Baseline to immediately and 2-months Post-Treatment.
  Evaluation of treatment differences (active versus sham) in change in Digit Span Forward & Backward. Metric: Memory Span
Rey-Osterrieth Complex Figure Test | Treatment differences (active versus sham) in change from Baseline to immediately and 2-months Post-Treatment.
  Evaluation of treatment differences (active versus sham) in change in Rey-Osterrieth Complex Figure Test scores. Metric: Score
The Digit Symbol Substitution Test | Treatment differences (active versus sham) in change from Baseline to immediately and 2-months Post-Treatment.
  Evaluation of treatment differences (active versus sham) in change on the Digit Symbol Substitution Test. Metric: Number of Items
Task-based electroencephalography (EEG) markers during a Go-NoGo task | Treatment differences (active versus sham) in change from Baseline to immediately and 2-months Post-Treatment.
  Evaluation of treatment differences (active versus sham) in EEG change on a Go-NoGo task with different levels of perceptual/semantic complexity. Metric: event-related potentials and time frequency changes.
Task-based electroencephalography (EEG) markers during a Semantic Object Memory Retrieval task | Treatment differences (active versus sham) in change from Baseline to immediately and 2-months Post-Treatment.
  Evaluation of treatment differences (active versus sham) in EEG change on a Semantic Object Retrieval task. Metric: event-related potentials and time frequency changes.

CONTACTS AND LOCATIONS:
Overall Officials: Hsueh-Sheng Chiang, MD, PhD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) will be shared in a de-identified format in accordance with NIH data-sharing policies and institutional guidelines.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available after publication of primary results or 12 months following study completion, whichever occurs first. The data will be accessible for at least 5 years post-publication.
Access Criteria: Qualified researchers may request access by submitting a data request with a description of the intended use.